CLINICAL TRIAL: NCT04955769
Title: Investigation of Body Image, Self-stigma, Intuitive Eating and Exercise Behavior in Overweight and Obese
Brief Title: Body Image, Self-stigma, Intuitive Eating and Exercise Behavior in Overweight and Obese
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nur Elcin Boyacıoglu, Assist. Prof, Istanbul University - Cerrahpasa
Other Study IDs: IstanbulUC9325
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Overweight and Obesity
Keywords: Intuitive Eating; Body Image; Self-Stigma; Exercise Behavior; Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study, it was aimed to investigate the relationship between body image, self-stigma, intuitive eating and exercise attitude levels, which are thought to be effective on the mental well-being of overweight and obese individuals. For this purpose, the Body Image Scale, Intuitive Eating Scale-2, Exercise Stages of Change Scale-Short Form and Decisional Balance Scale in Exercise will be used to assess overweight and obese individuals. 100 people will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18-65
* BMI ≥30 kg/m2,
* No surgical operation in the last 6 months

Exclusion Criteria:

* Musculoskeletal disorders or systemic diseases that may prevent exercise
* The presence of psychiatric or neurological disease affecting cooperation and cognitive functions
* Presence of acute pain
* Heart pain
* Presence of previous myocardial infarction, subjective heart failure, uncontrolled diabetes and hypertension

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Overweight and obese individuals between the ages of 18-65 will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Body Image Scale | Baseline
  It was developed by Secord and Jourand in 1953, and was adapted to Turkish society after being validated and reliable by Hovardaoğlu in 1989. The scale includes 40 items and each item is related to an organ or a part of the body (such as arm, leg, face) or a function (such as sexual activity level).
Intuitive Eating Scale-2 | Baseline
  The Intuitive Eating Scale-2 was developed by Tylka and Kroon Van Diest (2013) to measure intuitive eating behaviors. The scale consists of 21 questions and four sub-titles.

SECONDARY OUTCOMES:
Exercise Stages of Change Scale-Short Form | Baseline
  This 5-optioned scale evaluates the changes of exercise behavior of participants in five stages of pre contemplation, contemplation, preparation, action, and consistency. Participants have to select one of the 5 options that evaluate the intention to participate in physical activity and sports now and in the future.
Decisional Balance Scale in Exercise | Baseline
  The scale is used to measure the individual decision to exercise with 10 questions designed to evaluate exercise beliefs (positive beliefs and obstacles). Participants are asked to choose on a 5-point Likert scale, in what way important every statement was with respect to their intentions to exercise, or not.

CONTACTS AND LOCATIONS:
Overall Officials: Nur Elçin Boyacıoğlu, Assist Prof, Principal Investigator — Istanbul Universitesi-Cerrahpasa
Locations (1):
- DiyeTat-Beslenme ve Danışmanlık, Istanbul, Kadıköy, Turkey (Türkiye)